CLINICAL TRIAL: NCT00674960
Title: Phase 1 Study to Determine the Efficacy of Using Far Infrared Radiation for the Management, Control and Treatment of Frontotemporal Dementia (Pick's Disease)
Brief Title: Far Infrared Irradiation for the Management, Control and Treatment of Frontotemporal Dementia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: : Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-FD-CTP1
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Pick Disease of the Brain
Keywords: Brain Atrophy, Circumscribed Lobar; Circumscribed Lobar Atrophy of the Brain; Lobar Atrophy (Brain); Pick Disease; Pick's Disease; Picks Disease of Brain
MeSH Terms: conditions — Pick Disease of the Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Radiation: Far Infrared Radiation (5μm to 20μm wavelength)
  Interventions: Radiation: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)

INTERVENTIONS:
Radiation: Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Far Infrared Radiation (5μm to 20μm wavelength). Far Infrared radiation for 30 to 40 minutes per treatment session.
  Other Names: Far Infrared Radiation (5μm to 20μm wavelength)

SUMMARY:
Pick's disease, also known as Pick disease,or FTD is a rare fronto-temporal neurodegenerative disease. This study will investigate the use of far infrared radiation for the control, management and treatment of Pick's disease.

DETAILED DESCRIPTION:
This disorder causes progressive destruction of nerve cells in the brain and causes tau proteins to accumulate into the "Pick bodies" that are a defining characteristic of the disease. Tau proteins are microtubule-associated proteins that are abundant in neurons in the central nervous system and are less common elsewhere.

Observations from our research studies indicate that, far infrared rays provide energy to the body, improve the autonomic functions of the nervous system, restore the functions of the endocrine system, strengthen the immune system, improve blood circulation and increase the level of oxygen in the cells and promote the regeneration of muscle cells, nerves and brain cells.

It is hereby postulated that irradiation using far infrared, with wavelength between 5 to 20 microns, of the central nervous system, the endocrine system and the whole body could prevent, control, manage or possibly lead to complete rehabilitation of people who have FTD.

ELIGIBILITY:
Inclusion Criteria:

* People with Pick's Disease

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Therapy for FTD patients | 1 year

SECONDARY OUTCOMES:
Rehabilitation of FTD Patients | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada